CLINICAL TRIAL: NCT01431586
Title: A Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single, Escalating Oral Doses of JDTic in Healthy Male Subjects
Brief Title: First in Humans Study of JDTic
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No further subjects will be enrolled due to adverse events.
Sponsor: RTI International (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: JDTic-001; U19DA021002 (NIH)
Record Dates: First submitted 2011-08-31; First posted 2011-09-09 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Cocaine Dependence
Keywords: JDTic; cocaine dependence; kappa-opioid antagonist
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single dose JDTic 1 mg, 3 mg, or 10 mg (Experimental)
  Interventions: Drug: JDtic

INTERVENTIONS:
Drug: JDtic — The planned JDTic dose levels to be evaluated are 1 mg, 3 mg, and 10 mg; however, the actual dose levels evaluated may be different, and/or additional dose levels may be added by protocol amendment, depending on the safety and PK results of the lower doses.
  Subjects will be admitted to the clinic the day before dosing and will be confined to the clinic for 6 nights, with safety and PK evaluations and assessments lasting approximately 125 hours following administration of study drug.

SUMMARY:
This is the first study to be conducted in humans for JDTic, a new chemical entity, with evaluations focusing on the safety, tolerability, and pharmacokinetics (PK) of JDTic following administration of single oral doses. JDTic is a novel, selective κ opioid receptor antagonist and is currently being developed by RTI International as a potential pharmacotherapy to treat cocaine dependence. This study has the possibility of identifying the maximum tolerated dose in humans and a surrogate measure of JDTic pharmacodynamic (PD) activity. Data from this study will be used to plan for and define dose ranges for subsequent studies, as well as to identify potential indicators of JDTic pharmacological activity.

DETAILED DESCRIPTION:
JDTic-001 will be a single-center, double-blind, placebo-controlled, single-dose study evaluating three planned escalating oral doses of JDTic in three planned cohorts of healthy male subjects without a history of illicit drug use within the 12 months preceding the Screening Visit, or other substances of abuse within the 12 months preceding the Screening Visit. Each cohort of up to 8 eligible subjects will be enrolled sequentially to receive a single oral dose of study drug under fasting conditions. JDTic dose escalation will occur only if safety and PK data permit. A semi adaptive dosing plan will be followed such that the first two dose cohorts will comprise 4 subjects each and the third planned cohort will comprise 8 subjects. If adverse events (AEs) considered to be at least possibly related to study medication by the Clinic Principal Investigator are noted in study subjects participating in the first two cohorts, an additional 4 subjects will be dosed at the same dose level as part of the affected cohort, unless otherwise determined by the Safety Review Team (SRT) as guided by the JDTic-001 Data and Safety Monitoring Plan (DSMP). Should dosing of additional subjects occur in the first cohort of subjects, then the second cohort of subjects will also include 8 subjects. In each cohort, subjects will be randomized 3:1 active drug: placebo in a double-blind fashion.

The planned JDTic dose levels to be evaluated are 1 mg, 3 mg, and 10 mg; however, the actual dose levels evaluated may be different, and/or additional dose levels may be added by protocol amendment, depending on the safety and PK results of the lower doses.

Subjects will be admitted to the clinic the day before dosing and will be confined to the clinic for 6 nights, with safety and PK evaluations and assessments lasting approximately 125 hours following administration of study drug. Subjects will be required to remain confined to the clinic for more than 6 nights if they experience persistent AEs that require observation and/or the Clinic Principal Investigator or qualified designee (physician who is listed as a subinvestigator on FDA Form 1572) considers it unsafe to release the subject from the clinic. Additionally, alternate subjects admitted with Group 1 but not dosed may remain in the clinic overnight for the possibility of being dosed with Group 2 and therefore would spend more than 6 nights in the clinic. Subjects will return to the clinic at 14 days after receiving their dose for a follow-up visit. If, at this visit, changes in the POMS™ assessment are noted that are considered significant in the Clinic Principal Investigator's opinion, or if a subject has an ongoing AE, the subject will return to the clinic every 14 days (or sooner, if clinically indicated) from the date of the follow-up visit until these changes/AEs have resolved. Subject participation in the study will last up to 4 weeks, from screening through the follow-up visit, depending on the date the subject's screening visit begins with respect to the date he is dosed, and provided no additional follow-up visits are necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Subject provides signed and dated, written informed consent before any study-specific procedures are performed, including washout of any medications. Subjects will be asked to meet the food, beverage and physical activity restrictions required for the screening visit prior to signing consent.
2. Subject is a healthy adult male aged 18 to 50 years, inclusive, at the time of consent.
3. Subject has a body weight of at least 50 kg and a body mass index (BMI) in the range of 18 to 30
4. Subject has a negative prestudy urine drug screen and no history of use of illicit drugs within 12 months of the screening visit or other substances of abuse within 12 months of the screening visit.
5. Subject has not used tobacco for at least 90 days prior to screening.
6. Subject has no history of any cardiovascular disease and no clinically significant ECG results at screening.
7. Subject is negative for hepatitis C (HCV) antibodies, hepatitis B (HBV) surface antigen, and human immunodeficiency virus (HIV) at screening.
8. Subject is in good general health in the opinion of the Clinic Principal Investigator and as determined by medical history, physical examination, orthostatic vital signs (supine, sitting, and standing blood pressure and heart rate; supine respiratory rate and oral temperature), 12-lead ECG, and clinical laboratory tests at screening. Additionally, the subject's clinical laboratory test results must meet the following criteria:

   - Within normal limits: Reticulocyte count

   - Within upper limit of normal and not clinically significantly below the lower limit of normal: Aspartate aminotransferase (AST) Alanine aminotransferase (ALT) Gamma glutamyl transferase (GGT) Prothrombin time (PT) Activated partial thromboplastin time (aPTT) Serum troponin I Blood urea nitrogen (BUN) Creatinine Bilirubin, total Alkaline phosphatase Creatine kinase Lactate dehydrogenase (LDH)

   - No clinically significant abnormalities: Sodium Protein, total Calcium Chloride Phosphorus Albumin Globulin Cholesterol Triglycerides Red blood cells (RBC) White blood cells (WBC) Hematocrit Hemoglobin Platelets Glucose Potassium WBC differential RBC indices Uric acid Urinalysis
9. Subject is willing to use barrier contraception with spermicide during sexual intercourse and is also willing to not donate sperm while enrolled in this study and for at least 90 days after receiving his dose of study drug.
10. Subject is willing and able to comply with study instructions and restrictions and is available to complete the study assessments as required by the protocol
11. Subject is fluent in English.

Exclusion Criteria:

1. Subject has a history or evidence of hepatic, GI, renal, respiratory, ophthalmic, cardiovascular, hematologic, endocrine/metabolic, neurologic, immunologic, oncologic, or psychiatric illness or significant abnormalities; OR other condition(s)/surgical intervention(s) known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
2. Subject has a clinically significant abnormal ECG at screening or prior to dosing. Multiple premature atrial contractions or multiple premature ventricular contractions (PVCs), with the exception of non-clinically significant unifocal PVCs, are considered clinically significant, as are bundle branch blocks, second or third degree heart block, or any arrhythmia other than respiratory sinus arrhythmia.
3. Subject has one or more ECG parameters outside the following ranges at Screening or just prior to dosing:

   Heart rate less than 55 or greater than 100 beats per minute (bpm), PR interval less than 120 or greater than 180 msec, QRS duration less than 70 or greater than 100 msec, QT interval (Bazett) greater than 420 msec
4. One or more of the Subject's supine vital signs are outside the ranges specified below:

   * Systolic blood pressure: 90-140 mmHg, inclusive
   * Diastolic blood pressure: 60-90 mmHg, inclusive
   * Heart rate: 55-100 beats per minute (bpm), inclusive
   * Respiratory rate: 12-20 breaths per minute, inclusive
   * Oral temperature: 97.0-99.7 degrees Fahrenheit, inclusive
5. Subject has a history or current evidence of early cardiac repolarization.
6. Subject has a history or family history of QT prolongation, arrhythmia, or uncontrolled hypertension.
7. Subject has a history of seizure, head injury, neurosurgery or brain trauma, or a family history of nontraumatic seizure.
8. Subject has an infection of any type or clinically significant abnormality identified by the screening medical or laboratory evaluations.
9. Subject has consumed alcohol within 48 hours prior to the screening visit or is unwilling to discontinue alcohol consumption within 48 hours of being admitted to the clinic.
10. Subject has a history of significant alcohol consumption, defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units, with 1 unit equivalent to 1 can or bottle (12 oz) of beer, or 1 measure (1.5 oz) of spirits, or 1 glass (5 oz) of wine.
11. Subject is unwilling to discontinue the consumption of caffeine containing beverages 72 hours prior to clinic admission.
12. Subject has consumed or is unwilling to abstain from consuming grapefruit or grapefruit-, poppy seed-, or quinine-containing substances, within 14 days of clinic admission.
13. Subject has used a prescription medication within 30 days prior to receiving his dose of study medication; or has used nonprescription medications, dietary supplements, or herbal supplements within 14 days of receiving his dose of study medication, with the exception of acetaminophen, which may be taken up to 24 hours prior to dosing.
14. Subject has had any acute GI illness or infection within 14 days prior to receiving his dose of study medication.
15. Subject has participated in an investigational trial within 45 days prior to receiving his first dose of study medication.
16. Subject is unable to donate blood, has a clotting disorder(s), or has donated blood or lost a significant amount of blood within 8 weeks prior to screening.
17. Subject has an unexplained weight loss or gain (greater than 10 percent) within 30 days prior to screening.
18. Subject has an allergy to or has experienced side effects with opioid antagonists
19. Subject is unable to respond to or recognize potential side effects of the study drug. This may include, but is not limited to, subjects with a mental illness or disorder.
20. Subject has any condition or set of circumstances not otherwise excluded that in the judgment of the Clinic Principal Investigator could interfere with the subject's ability to comply with the protocol requirements and restrictions and completion of study evaluations, or could pose safety risks to the subject.
21. Subject has performed strenuous exercise within 48 hours prior to the screening examination or refuses to abstain from strenuous exercise from the date of consent provision until the completion of the follow-up visit.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single, escalating oral doses of JDTic in healthy male subjects | 125 hours following administration of JDTic
  Safety and tolerability of JDTic: clinical signs and symptoms, adverse events (AEs), vital signs, electrocardiographic parameters, clinical laboratory test results, psychomotor function assessment

SECONDARY OUTCOMES:
Pharmacokinetics Profile | 125 hours post-dose
  PK parameters of JDTic: maximum concentration (Cmax), time to maximum concentration (tmax), area under the curve from time zero to last timepoint with measurable concentration, area under the curve from time zero to infinity, terminal elimination half-life (t1/2) and corresponding elimination rate constant, apparent total body clearance (CL/F), and amount excreted in urine (Aeurine)
To evaluate a potential surrogate measure of JDTic PD activity | 14 days after receiving JDTic
  Exploratory pharmacologic activity measure of JDTic: Profile of Mood States™ (POMS™)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Swearingen, MD, Principal Investigator — Celerion
Locations (1):
- Celerion Inc., Tempe, Arizona, United States